CLINICAL TRIAL: NCT00868036
Title: Contact Allergens Causing Chronic Urticaria in a New England-Area Population
Brief Title: Evaluating for Contact Allergies in Patients With Chronic Urticaria
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: American Contact Dermatitis Society (ACDS) (Other)
Responsible Party: Sponsor
Other Study IDs: Contact Urticaria; IRB #8343; ACDS (Other Grant/Funding Number: American Contact Dermatitis Society)
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Urticaria; Patch Testing; Dermatitis; Allergy; Contact Sensitization
Keywords: urticaria; hives; dermatitis; rash; contact dermatitis; contact; contact sensitization; allergy; allergen; patch testing; IgG; delayed-hypersensitivity reaction; hypersensitivity
MeSH Terms: conditions — Urticaria; Dermatitis; Hypersensitivity; Exanthema; Dermatitis, Contact; Hypersensitivity, Delayed | interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patch testing: Patch testing on patients with chronic idiopathic dermatitis.
  Interventions: Procedure: Patch Testing

INTERVENTIONS:
Procedure: Patch Testing — Patch testing will be performed with a modified North American Contact Dermatitis Group (NACDG) standard series, cosmetics/preservative, fragrance, and textile series in all patients. Based on patient history, other appropriate allergen series will be added. After two days, patches will be removed and the areas will be inspected for type IV hypersensitivity reactions including papules, edema or vesicles.
  Results will be graded and interpreted at a "delayed read," 3-4 days after allergens are placed with patch testing.
  Other Names: North American Contact Dermatitis Group (NACDG)

SUMMARY:
Hives affects 10-25% of the population worldwide at some time during their lifetime. Hives are itchy transient swellings of the skin lasting 4-36 hours. Chronic urticaria is defined as hives that have been ongoing for six weeks or more.

Patch testing is performed to diagnose allergic contact dermatitis, and if contact allergens are found via patch testing, patients can often be cured of their dermatitis. However, patch testing is currently not routinely performed in the evaluation of patients with chronic idiopathic urticaria.

Our hypothesis is to see if contact allergens can be identified with patch testing in patients with chronic urticaria, and, if any allergens are identified, to see if avoiding these contact allergens will make the chronic urticaria go away.

DETAILED DESCRIPTION:
Study Visits: Patients will be seen on Day #0, which will be a Monday, and the study will be explained. If they agree to participate, consent will be signed and they will be interviewed to determine any relevant occupational or personal exposures to potential allergens. They will be examined to determine if they have sufficient normal skin to undergo patch testing. Patients will be allowed to use antihistamines to treat pruritus as antihistamines do not abrogate T-cell-mediated immune reactions.

Scanpor (paper) tape strips of 10 allergens each contained within 10-mm Finn (aluminum) chambers will be applied to the patient's back. All patients will be tested to the Tufts Medical Center standard series, fragrance, cosmetics/preservative, and textile series. Based on patient history, other appropriate allergen series will be added.

After two days (on Day #2, a Wednesday), patches will be removed and the areas will be inspected for type IV hypersensitivity reactions including papules, edema or vesicles. The testing areas will be marked using a surgical marker and the patients will return the following day (on Day #3, a Thursday) for a delayed reading.

Interpretation: Patch test reactions will be interpreted by using NACDG criteria: negative reaction (macular erythema); 1+ (weak reaction; non-vesicular erythema, infiltration, and possibly papules); 2+ (strong reaction; edematous or vesicular); 3+ (extreme reaction; spreading, bullous, or ulcerative lesions), or irritant reaction. If contact allergens are found, patients will be educated about allergen avoidance and given listings from the Contact Allergen Replacement Database delineating products they may use which do not contain their allergens.

Follow-up Interview: One to three months after patch testing, the patients will be contacted to determine whether allergen avoidance has resulted in any improvement in their chronic urticaria. They will be asked how well they have adhered to allergen avoidance (completely avoided, mostly avoided, somewhat avoided, or not at all avoided) and how their urticaria has been since changing their habits (a response score: completely resolved, mostly improved, somewhat improved, no change, or worse).

Costs: there will be no costs to the patients to participate in this study. Patients will be seen as regular patients at Tufts Medical Center, and their insurance providers will be billed for the visits. A stipend will be provided to patients to cover the costs of their transportation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a documented diagnosis of chronic urticaria, which is defined as:

  * urticaria (hives), in which each individual lesion lasts less than 48 hours,
  * urticaria which occurs several times per week,
  * urticaria which has lasted in this manner for a minimum of 6 weeks.

Referring physicians will be asked to provide this documentation, and patients will be asked to confirm these characteristics. Patients should have already undergone a workup to exclude other causes of their urticaria, and if any abnormalities have been encountered, these abnormalities would need to be insufficient to explain the extent of their urticaria.

Exclusion Criteria:

* Those patients with an explanation for their chronic urticaria.
* Patients may have their test postponed if they are currently using topical steroids to the area to be tested, or are taking prednisone or its equivalent daily.

Due to PI moving locations, no additional information available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Due to PI moving locations, information not available.
Enrollment: 23 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
PI changed location, no additional information available. To identify contact allergens with patch testing in patients with chronic idiopathic urticaria living in the New England area. | Late read: three days after allergens for patch testing are placed

SECONDARY OUTCOMES:
PI changed location, no additional information available. To determine if avoidance of contact allergens causes the resolution of chronic urticaria in those patients with positive patch test results. | 1-3 months after patch testing performed.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Scheinman, M.D., Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

REFERENCES:
- [Background] Guerra L, Rogkakou A, Massacane P, Gamalero C, Compalati E, Zanella C, Scordamaglia A, Canonica WG, Passalacqua G. Role of contact sensitization in chronic urticaria. J Am Acad Dermatol. 2007 Jan;56(1):88-90. doi: 10.1016/j.jaad.2006.07.023. Epub 2006 Oct 20. PMID 17190624
- [Background] Wai YC, Sussman GL. Evaluating chronic urticaria patients for allergies, infections, or autoimmune disorders. Clin Rev Allergy Immunol. 2002 Oct;23(2):185-93. doi: 10.1385/CRIAI:23:2:185. PMID 12221863